CLINICAL TRIAL: NCT03581734
Title: Study on the Immunogenicity of Oral Polio Vaccine (OPV) and Oral Cholera Vaccine (OCV) When Co-administered
Brief Title: Immunogenicity of Co-administered Oral Polio Vaccine and Oral Cholera Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-17120
Record Dates: First submitted 2018-06-25; First posted 2018-07-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Vaccine Reaction
Keywords: Oral Polio Vaccine; Oral Cholera Vaccine; Co-administration; Immunogenecity
MeSH Terms: interventions — Poliovirus Vaccine, Oral; Cholera Vaccines

STUDY DESIGN:
Intervention Model Description: We propose to conduct an open-label, randomized controlled study in Dhaka, Bangladesh, among healthy children aged 1 - 3 years old who have received either no dose or one dose of OPV and has not received any dose of IPV or OCV at any time before enrolment based upon immunization card record or history from parents after full informed consent. Participants will be randomized to one of three groups ; (i) OPV only, (ii) OCV only, or (iii) co-administered OPV and OCV
Who Masked: Outcomes Assessor
Masking Description: Laboratory staff will remain blinded throughout the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- OPV only (Active Comparator): The vaccine will be available in prefilled vials containing 10 doses. Each vial will be labelled with the study ID of the participant. Therefore, for participants randomized to arm A and arm C, there will be 3 vials per participant for the 3 doses of the bOPV vaccine to be given 28 weeks apart. Any remaining, non-used doses of vaccine in the vial will be discarded.
  Interventions: Biological: Oral Polio Vaccine
- Shanchol only (Active Comparator): Each dose of vaccine is 1.5ml in volume. Each vial will be labelled with the study ID of the participant. One vial will be used per participant per study visit. OCV was studied in a double-blind, randomized, placebo-controlled trial in Kolkata, India. Participants were 1 year and above in age. In these studies, 100 children aged 1-17 were administered 2-doses of OCV or placebo separated by an interval of two weeks, with 80% of vaccinated showing over 4 fold rise in serum V. cholerae O1 antibody titers, showing that the 2-dose regimen was well-tolerated, safe and immunogenic
  Interventions: Biological: Oral Cholera Vaccine
- OPV-OCV co-administered (Experimental): Our primary analysis will be to compare seroconversion (defined as a change of status from seronegative to seropositive titers, or a ≥4-fold rise in antibody titer) for OPV1 and OPV 3 antibodies between Arm A and Arm C, to determine whether seroconversion to bOPV when administered with Shanchol is non-inferior to seroconversion to bOPV when bOPV is administered alone.
  Our second objective will be to compare vibriocidal antibody seroconversion (also, ≥4-fold rise in antibody titers) to Shanchol when co-administered with OPV or when Shanchol is administered alone, Arm B compared to Arm C
  Interventions: Biological: Oral Polio Vaccine; Biological: Oral Cholera Vaccine

INTERVENTIONS:
Biological: Oral Polio Vaccine — OPV is a mixture of live attenuated poliovirus strains of each of the three serotypes, selected by their ability to mimic the immune response following infection with wild polioviruses, but with a significantly reduced incidence of spreading to the central nervous system.
  Arms: OPV only; OPV-OCV co-administered
Biological: Oral Cholera Vaccine — Bivalent, Killed, Whole Cell Oral Cholera Vaccine
  Arms: OPV-OCV co-administered; Shanchol only

SUMMARY:
Concomitant administration of multiple vaccines, including live attenuated immunizations, is safe and effective. Some restrictions apply for live vaccines; administering a live-virus vaccine within 4 weeks after administration of another live-virus vaccine can decrease immunogenicity to the second administered vaccine. Thus, it is recommended that live-virus vaccines should be administered the same day or ≥4 weeks apart. Data on co-administration of the currently available whole-cell killed Oral Cholera Vaccine (OCVs) with other oral vaccines, specifically, oral polio vaccines (OPV) is lacking. Although the risk of immunological interference due to co-administration of live vaccines with non-live vaccines is considered small if at all, a theoretical concern of interference has been raised. Given the substantial geographic correlation between polio- and cholera-affected and at-risk areas, which include some of the world's most impoverished and hard-to-reach populations, a strategy of co-administration of OCV with OPV to children targeted to receive OPVs has the potential to optimize the use of limited resources and improve coverage for both vaccines. The manufacturer recommendation for a two-week interval between administration of OPV and OCV precludes an integrated campaign or routine use in which OCV could be co-administered with OPV.

DETAILED DESCRIPTION:
Objectives of the study:

Primary :

1. To compare seroconversion for OPV types P1 and P3 when administered alone versus when administered with OCV on day 28 and 56 after vaccination.
2. To compare vibriocidal antibody response (based on a ≥ 4-fold rise) to OCV when administered alone versus when co-administered with OPV on day 28 and day 56 after vaccination.

   Secondary:
3. To determine safety of co-administration of OPV with OCV compared to OPV or OCV alone.

Hypothesis:

Co-administration of oral polio vaccine (OPV) and oral cholera vaccine (OCV) will not decrease immunogenicity of either vaccine among children 1 - 3 years old.

Research Design and Methods :

We propose to conduct an open-label, randomized controlled study in Dhaka, Bangladesh, among healthy children aged 1 - 3 years old who have received either no dose or only one dose of OPV ( 0 - 1 dose) and has not received any dose of IPV or OCV at any time before enrolment based upon immunization card record or history from parents after full informed consent. Participants will be randomized to one of three groups ; (i) OPV only, (ii) OCV only, or (iii) co-administered OPV and OCV.

Schedule and description of observations and visits:

Participants will be randomized to one of three arms. First one is OPV only group, second one is OCV only and the last arm is Co-administration of OPV and OCV group. Each arm contains same number of participants (193). In each arm there will be three visits and blood collection. In case of OPV only group visit 1 will be considered as Day 0, Visit 2 will be considered as Day 28 (range 25th to 35th Day) and Visit 3 will be considered as Day 56 (range 50th to 70th Day).

In case of Shanchol only group visit, 1 will be considered as Day 0, Visit 2 will be considered as Day 28 (range 25th to 35th Day). As this participant misses his/her OPV, the plan has been taken to vaccinate them with OPV. For these children visit 3 will be considered as Day 56 (range 50th to 70th Day) and will get OPV only. For catch up, doses Visit 4 will be considered as Day 84 (range 75th to 105th) and Visit 5 will be considered as Day 112 (range 100th to 140th Day) and will get bivalent oral polio vaccine (bOPV) and inactivated polio vaccine (IPV).

In case Co-administration of OPV and OCV group, visit 1 will be considered as Day 0, Visit 2 will be considered as Day 28 (range 25th to 35th Day). Participants will get bOPV and Shanchol simultaneously in these 2 different day visits. Visit 3 will be considered as Day 56 (range 50th to 70th Day) and will get bOPV and IPV.

Study Area Recruitment will occur in urban slums in Hazaribagh, Kamrangirchar and Rayerbazar in Southern Dhaka.

Inclusion criteria

* Apparently healthy children aged 1 to 3 years of age.
* Family able to understand and comply with planned study procedures and consents to be in the study
* Have received either no dose or only one dose of OPV ( 0 - 1 dose) and has not received any dose of IPV or OCV at any time before enrollment based upon immunization card record or history from parents.

Exclusion criteria:

* Parents and children who are unable/unwilling to participate in the full length of the study for any reason.
* Child/family planning on moving away from the study area during the study period
* A diagnosis, suspicion of, or clinical condition consistent with an immunodeficiency disorder (either in the child or in a member of the immediate family).
* A suspicion or known history of bleeding disorder that would contraindicate venipuncture.
* Acute diarrhea, infection or illness at the time of the first visit that would require the child's admission to a hospital or would contraindicate provision of OPV per country guidelines.
* History of severe allergic reaction to a component of the study vaccine
* Acute vomiting or diarrhea within 24 hours before the first visit.
* Severely malnourished children( Z score <-3 )
* Previously received 3 doses of OPV or a single dose of IPV or OCV at any time before enrollment based upon immunization card record.

Study Intervention

Description of vaccines Three different vaccines will be used in this study: bOPV, IPV and OCV.

1. Bivalent oral polio vaccine (bOPV)
2. Inactivated polio vaccine (IPV)
3. Inactivated Oral cholera vaccine (OCV)

Outcome measures/variables:

Primary

1. Anti-poliovirus antibodies type 1 and type 3 microneutralization titer when OPV and OCV are administered separately, and when given together.
2. Vibriocidal antibody response to V. cholerae O1, serotype Ogawa and Inaba when OPV and OCV are administered separately and when given together.

Secondary

1. Number of adverse events and serious adverse events between OPV and OCV when given alone versus when given concomitantly.

Assessment after vaccination

Monitoring for adverse events After administration of each vaccine dose, all study participants will be observed for 30 minutes to monitor for potential allergic reactions to the vaccine. A short interview will also be conducted to identify if side effects including diarrhea (3 or more loose stools over 24 hours), nausea, vomiting or rash were experienced with prior vaccine administration. For OCV recipients, the participant adverse event follow-up period will be 14 days after each dose. For OPV and IPV adverse event follow up will be 30 minutes after receiving the vaccine, as per national guidelines.

Reporting Procedures for Serious Adverse Events (SAEs):

All SAEs that occur during the study will be reported by the study PI or designee within 24 hours of learning about the incident to the ethical review committee (ERC) and the data safety monitoring board (DSMB). The SAE form will always be completed as thoroughly as possible with all available details of the event, signed by the principal investigator. If the investigator does not have all the information regarding an SAE, he/she will not wait to receive additional information before submitting the report.

The study physicians/medical officers will follow-up the participants with SAEs until the event has: resolved, subsided, stabilized or disappeared or the event is otherwise explained, or the participant is lost to follow-up.

Data Collection and Management Procedures

Data management:

Study personnel will directly collect data through tabloid PC except for adverse event (AE) data. Adverse Event data will be collected in hard-copies and will be double-entered into computers in a dedicated area located at icddr,b, using data entry programs.

Methods for specimen collection, storage and processing

Specimen Collection:

Approximately 2-3 ml of blood will be collected before administration of the first study vaccine (Day 0), before the second study vaccine administration (Day 28) and before catch-up vaccine administration (Day 56).

Specimen Testing:

Sera collected before and after each of the 3 doses of study vaccines will be examined for the presence (detectable) or absence of neutralizing antibodies to all three poliovirus serotypes and to cholera following a standard protocol. Laboratory testing will be conducted to determine antibody responses to OPV at the Centers for Disease Control and Prevention (CDC), Atlanta and antibody response to OCV at icddr,b.

Specimen shipment To evaluate vaccine immunogenicity serum specimens will be processed at icddr,b's Mucosal Immunology & Vaccinology Laboratory. Research specimens collected for the immunogenicity time points will be separated into aliquots by the icddr,b Mucosal Immunology & Vaccinology Laboratory per study specific procedures and stored for immunological analysis and for potential shipment to the Enterovirus Laboratory at the Division of Viral Diseases, CDC in Atlanta, United States by following International Air Transport Association (IATA) guidelines.

Data Analysis The primary analysis will be to compare seroconversion (defined as a change of status from seronegative to seropositive titers, or a ≥4-fold rise in antibody titer) for OPV1 and OPV 3 antibodies between Arm A and Arm C, to determine whether seroconversion to bOPV, when administered with Shanchol, is non-inferior to seroconversion to bOPV when bOPV is administered alone.

The second objective will be to compare vibriocidal antibody seroconversion (also, the ≥4-fold rise in antibody titers) to Shanchol when co-administered with OPV or when Shanchol is administered alone, Arm B compared to Arm C Statistical Analysis Primary Analytical Approach The primary analytical approach will be an intention-to-treat (ITT) analysis, which will include all participants originally enrolled in the study.

Secondary Analytical Approach We will also perform a per-protocol (PP) analysis, which will include only those children who adhered to the study protocol (e.g. received all 3 planned vaccine doses at the adequate intervals ± 3 days and have testable blood samples).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children aged 1 to 3 years of age. Family able to understand and comply with planned study procedures and consents to be in the study.
* Have received either no dose or only one dose of OPV ( 0 - 1 dose) and has not received any dose of IPV or OCV at any time before enrollment based upon immunization card record or history from parents.

Exclusion Criteria:

* Parents and children who are unable / unwilling to participate in the full length of the study for any reason.
* Child / family planning on moving away from the study area during the study period
* A diagnosis, suspicion of, or clinical condition consistent with an immunodeficiency disorder (either in the child or in a member of the immediate family) or is on long-term (>3 months) of immunosuppressive therapy.
* A suspicion or known history of bleeding disorder that would contraindicate venipuncture.
* Acute diarrhea, infection or illness at the time of the first visit that would require the child's admission to a hospital or would contraindicate provision of OPV per country guidelines.
* History of severe allergic reaction to component of study vaccine
* Acute vomiting or diarrhea within 24 hours before the first visit.
* Severely malnourished children (Weight-for-age with z-score < - 3 below the median of the WHO child growth standards.)
* Previously received 3 doses of OPV or single dose of IPV or OCV at any time before enrollment based upon immunization card record.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 579 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-10-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
Anti-poliovirus antibodies | One year
  Anti-poliovirus antibodies P1 and P3 microneutralization titer when OPV and OCV are administered separately, and when given together.
Vibriocidal antibody response | One year
  Vibriocidal antibody response to V. cholerae O1, serotype Ogawa and Inaba when OPV and OCV are administered separately, and when given together.

SECONDARY OUTCOMES:
Safety: number of adverse events and serious adverse events | One year
  The number of adverse events and serious adverse events between OPV and OCV when given alone versus when given concomitantly.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Firdausi Qadri, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Hazaribagh Field Clinic, Dhaka, Bangladesh

REFERENCES:
- [Result] Patel M, Steele AD, Parashar UD. Influence of oral polio vaccines on performance of the monovalent and pentavalent rotavirus vaccines. Vaccine. 2012 Apr 27;30 Suppl 1:A30-5. doi: 10.1016/j.vaccine.2011.11.093. PMID 22520134
- [Result] Taniuchi M, Platts-Mills JA, Begum S, Uddin MJ, Sobuz SU, Liu J, Kirkpatrick BD, Colgate ER, Carmolli MP, Dickson DM, Nayak U, Haque R, Petri WA Jr, Houpt ER. Impact of enterovirus and other enteric pathogens on oral polio and rotavirus vaccine performance in Bangladeshi infants. Vaccine. 2016 Jun 8;34(27):3068-3075. doi: 10.1016/j.vaccine.2016.04.080. Epub 2016 May 3. PMID 27154394
- [Result] Emperador DM, Velasquez DE, Estivariz CF, Lopman B, Jiang B, Parashar U, Anand A, Zaman K. Interference of Monovalent, Bivalent, and Trivalent Oral Poliovirus Vaccines on Monovalent Rotavirus Vaccine Immunogenicity in Rural Bangladesh. Clin Infect Dis. 2016 Jan 15;62(2):150-6. doi: 10.1093/cid/civ807. Epub 2015 Sep 8. PMID 26349548
- [Derived] Islam MT, Date K, Khan AI, Bhuiyan TR, Khan ZH, Ahmed S, Hossain M, Khaton F, Zaman K, McMillan NAJ, Anand A, An Q, Zhang C, Weldon WC, Yu A, Luby S, Qadri F. Co-administration of Oral Cholera Vaccine With Oral Polio Vaccine Among Bangladeshi Young Children: A Randomized Controlled Open Label Trial to Assess Interference. Clin Infect Dis. 2023 Jan 13;76(2):263-270. doi: 10.1093/cid/ciac782. PMID 36136760